CLINICAL TRIAL: NCT03739463
Title: Pro-omega-3, Reduction of Inflammation and Modulation of Prematurity
Acronym: Pro-MEGA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université de Sherbrooke (Other)
Collaborators: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MP-31-2018-2496
Record Dates: First submitted 2018-10-22; First posted 2018-11-13 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-10

CONDITIONS: PPROM
Keywords: Pro-omega-3; Inflammation; Prematurity
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes; Inflammation; Premature Birth | interventions — docosahexaenoic acid monoacylglyceride; Oleic Acid; Sunflower Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAG-DHA (Experimental): 1500 MG of MAG-DHA per day until childbirth or for up to 2 weeks
  Interventions: Dietary Supplement: MAG-DHA
- Placebo (Placebo Comparator): 1500 MG of oleic acid per day until childbirth or for up to 2 weeks
  Interventions: Dietary Supplement: Oleic acid

INTERVENTIONS:
Dietary Supplement: MAG-DHA — 375 MG of MAG-DHA per capsules, two capsules BID
  Other Names: Pro-omega-3
  Arms: MAG-DHA
Dietary Supplement: Oleic acid — 375 MG of sunflower oil (oleic acid) per capsules, two capsules BID
  Other Names: Sunflower oil
  Arms: Placebo

SUMMARY:
The aim of the project is to decrease the inflammatory status of pregnant women with preterm premature rupture of membranes to delay the initiation of labour that would inevitably lead to premature delivery. The main objective is to measure the mean duration between the initiation of the treatment and delivery in the two groups treated either with MAG-DHA or with the placebo.

DETAILED DESCRIPTION:
This randomized controlled trial will be conducted in two hospitals in the province of Quebec (CHUS, CHUQ- Site mère-enfant Soleil).

Patients between 24 and 33 weeks of gestation with a diagnosis of preterm premature rupture of membranes (PPROM) who meet all inclusion and none of the exclusion criteria will be approached to participate. Once they have signed the IFC, participants will be randomized and begin a supplementation with either MAG-DHA or the placebo until delivery or for up to 2 weeks (14 days). A total of 70 patients will be recruited.

Principal outcome: To compare the difference in duration between the start of treatment and delivery between the group receiving MAG-DHA and the group receiving placebo.

Secondary outcomes: 1) Evaluate the difference in neonatal outcome between children in the MAG-DHA group and those in the placebo group. 2) Determine the inflammatory status of the patients associated with the exposure to either MAG-DHA or the placebo.

This regimen could potentially represent an innovative approach in the management of women with a diagnosis of PPROM.

ELIGIBILITY:
Inclusion Criteria:

* PPROM diagnosis, gestational age between 24 and 33 weeks of gestation.

Exclusion Criteria:

* multiple pregnancy, placenta previa, preeclampsia, retroplacental hematoma, chorioamnionitis, intrauterine growth retardation, severe fetal malformations

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnacy required
Enrollment: 70 (Estimated)
Dates: Start 2018-12-03 (Estimated); Primary Completion 2019-11-05 (Estimated); Study Completion 2020-05-15 (Estimated)

PRIMARY OUTCOMES:
Duration latency period | From PPROM through delivery

SECONDARY OUTCOMES:
Composite neonatal score | From birth through the first 28 days of life
  Composite neonatal score includes any one or more of the following: acute respiratory distress, bronchopulmonary dysplasia, proven sepsis, necrotizing enterocolitis, severe intraventricular hemorrhage (grade> 2) or periventricular leukomalacia
Inflammatory status | Every 2-3 days from PPROM until delivery or a maximum of 14 days, whichever happens first
  Inflammatory status will be determined based on the quantification of any one or more of the following biomarkers in blood and vaginal secretions specimens: resolvins, lipoxygenase isoforms

IPD SHARING:
Plan to Share IPD: Undecided